CLINICAL TRIAL: NCT03374137
Title: Post-Marketing Surveillance of Gazyva in Treatment of Patients With Gazyva in Follicular Lymphoma or Previously Untreated Chronic Lymphocytic Leukemia Patients
Brief Title: Observational Study to Monitor Safety and Effectiveness of Obinutuzumab in Follicular Lymphoma or Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30074
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Chronic Lymphocytic Leukemia; Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- obinutuzumab: Participants with follicular lymphoma or previously untreated chronic lymphocytic leukemia will be treated with obinutuzumab.
  Interventions: Biological: obinutuzumab

INTERVENTIONS:
Biological: obinutuzumab — Obinutuzumab 1000 mg solution used for infusion according to routine clinical practice.
  Other Names: Gazyva

SUMMARY:
This study aims to collect clinical data, mainly focused on safety, in the local target population as per the requirement of Korea Ministry of Food and Drug Safety for market authorization. The study population comprises patients with approved local indications chronic lymphocytic leukemia (CLL) and/or follicular lymphoma (FL) in routine clinical practice after launch.

ELIGIBILITY:
Inclusion Criteria:

* Administered obinutuzumab under the approved indications in Korea at investigator's discretion
* Previously untreated with obinutuzumab

Exclusion Criteria:

* Out-of locally approved indications, dosage, and administration
* Pregnant women, breastfeeding women
* Hepatic disease
* Participate in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants, who are going to receive obinutuzumab for one or more administrations according to medical opinions of the investigator in charge of surveillance, will be registered for this surveillance and treated with obinutuzumab under the approval conditions of the product in Korea
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Adverse Event (AE)/Adverse Drug Reaction (ADR) | from baseline until the end of the participant's observation period (up to approximately 8 years)
Percentage of Participants with Unexpected AE/ADR | from baseline until end of the participant's observation period (up to approximately 8 years)
Percentage of Participants with Expected ADR | from baseline until end of the participant's observation period (up to approximately 8 years)
Percentage of Participants with Non-serious ADR | from baseline until end of the participant's observation period (up to approximately 8 years)
Percentage of Participants with AEs of Special Interest (AESIs) | from baseline until end of the participant's observation period (up to approximately 8 years)

SECONDARY OUTCOMES:
Overall Response Rate | from baseline until end of the participant's observation period (up to approximately 8 years)
  According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 for CLL or Cheson 2014 criteria for FL
Stable Disease Rate | from baseline until end of the participant's observation period (up to approximately 8 years)
  According to IWCLL 2008 for CLL or Cheson 2014 criteria for FL
Progressive Disease Rate | from baseline until end of the participant's observation period (up to approximately 8 years)
  According to IWCLL 2008 for CLL or Cheson 2014 criteria for FL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- South Korea (17):
  - Inje University Busan Paik Hospital; Hematology-oncology, Busan
  - Pusan National University Hospital, Busan
  - St. Vincent's Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital; Department of Hematology, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Catholic Univ. of Incheon St.Mary's Hospital; Hemato-oncology, Incheon
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Borame Medical Center, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju